CLINICAL TRIAL: NCT00217698
Title: Multicenter Phase II Trial of Gefitinib (Iressa™) First Line Therapy Followed by Chemotherapy in Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Gefitinib as First-Line Therapy Followed by Gemcitabine and Cisplatin in Treating Patients With Stage III or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 19/03; EU-20519; ZENECA-AZ1839IL/0542 (Other: Pharmaceutical company)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; large cell lung cancer; squamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Cisplatin; Gefitinib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cisplatin
Drug: gefitinib
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Gefitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as gemcitabine and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Giving gefitinib as first-line therapy followed by gemcitabine and cisplatin after disease progression may be an effective treatment for non-small cell lung cancer.

PURPOSE: This phase II trial is studying how well gefitinib works as first-line therapy followed by gemcitabine and cisplatin in treating patients with stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of gefitinib as first-line therapy, in terms of response rate (complete and partial response) or stability of disease, in patients with de novo or recurrent stage IIIB or IV non-small cell lung cancer.

Secondary

* Determine the safety of this drug in these patients.
* Determine the efficacy of gemcitabine combined with cisplatin when administered after first-line gefitinib in these patients.
* Determine quality of life of patients treated with this regimen.

OUTLINE: This is an open-label, multicenter study.

Patients receive oral gefitinib once daily until disease progression or unacceptable toxicity. Within 3 weeks after documented disease progression, patients receive gemcitabine IV over 30 minutes on days 1 and 8 followed by cisplatin IV over 1 hour on day 1. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, weeks 3, 6, 12, 18, and then every 12 weeks thereafter during gefitinib treatment. During chemotherapy, quality of life is assessed 1 week prior to starting chemotherapy treatment, day 1 of courses 3 and 5, and then every 12 weeks until disease progression.

After completion of study therapy, patients are followed every 3 months.

PROJECTED ACCRUAL: 'A total of 24-63 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically* or cytologically* confirmed non-small cell lung cancer (NSCLC), including any of the following cellular subtypes:

  * Squamous cell carcinoma
  * Adenocarcinoma
  * Large cell carcinoma
  * Poorly differentiated NSCLC NOTE: *New biopsies or cytologic specimens required for primary resection specimens older than 2 years
* De novo or recurrent disease, meeting 1 of the following stage criteria:

  * Stage IIIB disease

    * Malignant pleural effusion OR supraclavicular node involvement (N3)
    * Not suitable for curative multimodal treatment or surgery
  * Stage IV disease
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan or MRI

  * Measurable lesion must be outside previously irradiated areas
* Immediate chemotherapy is not clinically mandatory
* No small cell lung cancer (SCLC) or SCLC combined with NSCLC
* No symptomatic and/or untreated brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10.0 g/dL

Hepatic

* Bilirubin normal
* AST or ALT ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN (5 times ULN in the presence of bone metastases)
* No unstable or uncompensated hepatic disease

Renal

* Creatinine clearance > 60 mL/min
* No unstable or uncompensated renal disease

Cardiovascular

* No unstable or uncompensated cardiac disease
* No myocardial infarction within the past 3 months

Pulmonary

* No clinically active interstitial lung disease

  * Asymptomatic patients with chronic stable radiographic changes allowed
* No unstable or uncompensated respiratory disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after completion of study treatment
* Able to swallow and retain oral medication
* No active infection
* No uncontrolled diabetes mellitus
* No history of allergic reactions or hypersensitivity attributed to compounds of similar chemical or biological composition to study drugs
* No other severe or uncontrolled systemic disease
* No other serious underlying medical condition that would preclude study participation
* No psychiatric disability that would preclude study compliance or giving informed consent
* No other malignancy within the past 5 years except adequately treated nonmelanoma skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Prior intrapleural or intrapericardial local chemotherapy allowed
* No prior chemotherapy for advanced disease
* More than 6 months since prior neoadjuvant or adjuvant systemic chemotherapy for NSCLC

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* Concurrent palliative radiotherapy allowed (except to brain metastases)

Surgery

* Not specified

Other

* No prior epidermal growth factor receptor-targeted therapy for NSCLC
* No concurrent use of any of the following CYP3A4 inducers:

  * Phenytoin
  * Carbamazepine
  * Rifampin
  * Barbiturates
  * Hypericum perforatum (St. John's wort)
* More than 30 days since prior participation in another clinical trial
* No other concurrent investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2003-11; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Disease stabilization (complete response [CR], partial response [PR], or stable disease [SD]) after 12 weeks of study treatment

SECONDARY OUTCOMES:
Disease stabilization (CR, PR, or SD) after 6 and 18 weeks of study treatment
Objective response (CR and PR) to gefitinib treatment after weeks 6, 12, and 18
Adverse reactions to gefitinib treatment measured after completion of study treatment
Time to progression (TTP) with gefitinib treatment after completion of study treatment
Event-free survival (EFS) with gefitinib treatment after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C. Betticher, MD, Study Chair — Insel Gruppe AG, University Hospital Bern
Locations (14):
- Switzerland (14):
  - Saint Claraspital AG, Basel
  - Universitaetsspital-Basel, Basel
  - Inselspital Bern, Bern
  - Kantonsspital Bruderholz, Bruderholz
  - Spitaeler Chur AG, Chur
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital, Liestal
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Regionalspital, Thun
  - Kantonsspital Winterthur, Winterthur
  - City Hospital Triemli, Zurich
  - Klinik Hirslanden, Zurich
  - UniversitaetsSpital Zuerich, Zurich

REFERENCES:
- [Result] D'Addario G, Rauch D, Stupp R, Pless M, Stahel R, Mach N, Jost L, Widmer L, Tapia C, Bihl M, Mayer M, Ribi K, Lerch S, Bubendorf L, Betticher DC. Multicenter phase II trial of gefitinib first-line therapy followed by chemotherapy in advanced non-small-cell lung cancer (NSCLC): SAKK protocol 19/03. Ann Oncol. 2008 Apr;19(4):739-45. doi: 10.1093/annonc/mdm564. Epub 2007 Dec 19. PMID 18096565